CLINICAL TRIAL: NCT05261126
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-0616 in Adults With Hypercholesterolemia
Brief Title: A Study of the Efficacy and Safety of Enclitide Chloride (MK-0616 Oral PCSK9 Inhibitor) in Adults With Hypercholesterolemia (MK-0616-008)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0616-008; MK-0616-008 (Other: MSD); jRCT2031210701 (Registry Identifier: jRCT); 2021-005221-24 (EudraCT Number)
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Hypercholesterolemia; Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — MK-0616

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Enclitide Chloride 6 mg (Experimental): Participants will receive 6 mg of enlicitide chloride orally QD for 8 weeks
  Interventions: Drug: Enclitide Chloride
- Enclitide Chloride 12 mg (Experimental): Participants will receive 12 mg of enlicitide chloride orally QD for 8 weeks
  Interventions: Drug: Enclitide Chloride
- Enclitide Chloride 18 mg (Experimental): Participants will receive 18 mg of enlicitide chloride orally QD for 8 weeks
  Interventions: Drug: Enclitide Chloride
- Enclitide Chloride 30 mg (Experimental): Participants will receive 30 mg of enlicitide chloride orally QD for 8 weeks
  Interventions: Drug: Enclitide Chloride
- Placebo (Placebo Comparator): Participants will receive enlicitide chloride-matching placebo orally QD for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enclitide Chloride — Enclitide Chloride administered orally
  Other Names: MK-0616
  Arms: Enclitide Chloride 12 mg; Enclitide Chloride 18 mg; Enclitide Chloride 30 mg; Enclitide Chloride 6 mg
Drug: Placebo — Placebo matching enclitide chloride administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of enclitide chloride, an oral PCSK9 inhibitor, in lowering low-density lipoprotein cholesterol (LDL-C) in participants with hypercholesterolemia. The primary hypothesis is that at least one of the four doses of enclitide chloride tested in this study is superior to placebo on percent change from baseline in LDL-C at Week 8.

ELIGIBILITY:
Inclusion Criteria:

* History of clinical atherosclerotic cardiovascular disease (ASCVD), or has an ASCVD risk equivalent and/or a 10-year risk of having an ASCVD event ≥5.0%, AND has a corresponding LDL-C that falls within the protocol-specified range at screening.
* Treatment with a stable dose of one or more lipid-lowering therapies for ≥30 days before screening, or has not received treatment with any lipid-lowering therapy for ≥30 days before screening.
* A female participant is not pregnant or breastfeeding, not a woman of child-bearing potential (WOCBP) or is a WOCBP and agrees to follow contraceptive guidance during the intervention period and for at least 8 weeks after the last dose of study intervention.

Exclusion Criteria:

* History of homozygous familial hypercholesterolemia (FH) based on genetic or clinical criteria.
* History of nephrotic syndrome.
* History of unstable angina, a myocardial infarction, percutaneous transluminal coronary angioplasty, transient ischemic attack, or stroke within 3 months before Screening.
* Has poorly controlled diabetes mellitus, defined as hemoglobin A1C (A1C) ≥9.0% at Screening.
* History of malignancy ≤3 years before screening, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, which have no timeframe limitations relative to screening.
* Currently participating in or has previously participated in an interventional clinical study within 3 months before Screening.
* Has moderate or greater renal insufficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (63):
- United States (20):
  - Westside Medical Associates of Los Angeles ( Site 0026), Beverly Hills, California
  - Clinical Trials Research ( Site 0007), Sacramento, California
  - National Research Institute (NRI) - Santa Ana ( Site 0024), Santa Ana, California
  - Excel Medical Clinical Trials ( Site 0042), Boca Raton, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0050), Coral Gables, Florida
  - ForCare Clinical Research ( Site 0017), Tampa, Florida
  - Healthcare Research Network - Chicago ( Site 0037), Flossmoor, Illinois
  - Midwest Institute For Clinical Research ( Site 0036), Indianapolis, Indiana
  - Cotton O'Neil Mulvane ( Site 0022), Topeka, Kansas
  - L-MARC Research Center ( Site 0003), Louisville, Kentucky
  - The University of Mississippi Medical Center-Clinical Research and Trials Unit ( Site 0028), Jackson, Mississippi
  - Jubilee Clinical Research ( Site 0047), Las Vegas, Nevada
  - New Mexico Clinical Research & Osteoporosis Center ( Site 0032), Albuquerque, New Mexico
  - Mid Hudson Medical Research ( Site 0004), New Windsor, New York
  - altoona center for clinical research ( Site 0045), Duncansville, Pennsylvania
  - Piedmont Research Partners ( Site 0005), Fort Mill, South Carolina
  - Dallas Diabetes Research Center ( Site 0012), Dallas, Texas
  - Center for Cardiometabolic Disease Prevention/Baylor College of Medicine ( Site 0051), Houston, Texas
  - Northeast Clinical Research of San Antonio ( Site 0014), San Antonio, Texas
  - National Clinical Research, Inc-research office ( Site 0019), Richmond, Virginia
- Germany (5):
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen ( Site 0504), München, Bavaria
  - Kardiologische Gemeinschaftspraxis ( Site 0502), Nuremberg, Bavaria
  - Ambulantes Herzzentrum Kassel ( Site 0501), Kassel, Hesse
  - Universitätsklinikum Leipzig ( Site 0500), Leipzig, Saxony
  - Charité Campus Virchow-Klinikum ( Site 0505), Berlin
- Japan (8):
  - Chubu Rosal Hospital ( Site 1612), Nagoya, Aichi-ken
  - Kyoto Okamoto Memorial Hospital ( Site 1611), Kuse-gun Kumiyama-cho, Kyoto
  - Kitada Clinic ( Site 1604), Osaka, Osaka
  - Medical Corporation Heishinkai OCROM Clinic ( Site 1600), Suita-shi, Osaka
  - Seiwa Clinic ( Site 1605), Adachi-ku, Tokyo
  - meiwa hospital ( Site 1602), Chiyoda-ku, Tokyo
  - Heishinkai Medical Group ToCROM Clinic ( Site 1601), Shinjuku-ku, Tokyo
  - Sekino Hospital ( Site 1603), Toshimaku, Tokyo
- Mexico (10):
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad-Endocrinology ( Site 0205), Guadalajara, Jalisco
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occident-Unidad de Investigación Clínica Cardio, Guadalajara, Jalisco
  - Bio Investigación AMARC, S.C. ( Site 0204), Mexico City, Mexico City
  - Hospital Angeles Mocel ( Site 0209), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0212), Mexico City, Mexico City
  - Unidad biomedica avanzada monterrey-Clinical Trials ( Site 0200), Monterrey, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares-Subinvestigation ( Site 0201), Ciudad Madero, Tamaulipas
  - Hospital Angeles Xalapa-Internal Medicine-Cardiology ( Site 0202), Xalapa, Veracruz
  - Medical Care and Research SA de CV ( Site 0211), Mérida, Yucatán
  - Centro de Atención e Investigación Clínica ( Site 0214), Aguascalientes
- Norway (8):
  - Akershus Universitetssykehus-Hjertemedisinsk Avdeling ( Site 0705), Lørenskog, Akershus
  - Nordlandssykehuset ( Site 0709), Bodø, Nordland
  - Stavanger Universitetssykehus ( Site 0706), Stavanger, Rogaland
  - Sykehuset i Vestfold-Hjerteseksjonen ( Site 0703), Tønsberg, Vestfold
  - Oslo Universitetssykehus Aker-Preventiv kardiologi Aker ( Site 0704), Oslo
  - Oslo Universitetssykehus Rikshospitalet-Kardiologisk avdeling ( Site 0702), Oslo
  - Oslo Universitetssykehus Ullevål-Hjertemedisinsk avdeling, Ullevål ( Site 0701), Oslo
  - Oslo Universitetssykehus Aker-Lipidklinikken ( Site 0700), Oslo
- South Korea (4):
  - Keimyung University Dongsan Hospital ( Site 1703), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 1702), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 1701), Seoul
  - Samsung Medical Center ( Site 1700), Seoul
- Turkey (Türkiye) (3):
  - Ege University Medicine of Faculty-Cardilogy Department ( Site 1003), Bornova, İzmir
  - Hacettepe Universitesi ( Site 1002), Ankara
  - Eskisehir Osmangazi University-Cardiology ( Site 1000), Eskişehir
- United Kingdom (5):
  - Royal Free Hospital ( Site 1311), London, England
  - Queen Elizabeth University Hospital-Glasgow Clinical Research Facility ( Site 1310), Glasgow, Glasgow City
  - Layton Medical Centre ( Site 1303), Blackpool, Lancashire
  - William Harvey Heart Centre ( Site 1308), London, London, City of
  - Walsall Manor Hospital ( Site 1309), West Midlands, Walsall

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ballantyne CM, Banka P, Mendez G, Garcia R, Rosenstock J, Rodgers A, Mendizabal G, Mitchel Y, Catapano AL. Phase 2b Randomized Trial of the Oral PCSK9 Inhibitor MK-0616. J Am Coll Cardiol. 2023 Apr 25;81(16):1553-1564. doi: 10.1016/j.jacc.2023.02.018. Epub 2023 Mar 6. PMID 36889610
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 668 participants screened for inclusion, 381 were randomized 1:1:1:1:1 to receive MK-0616 6 mg, 12 mg, 18 mg, 30 mg, or placebo. Of the 381 randomized participants, one participant did not receive at least one dose of study intervention.
Groups:
- MK-0616 6 mg: Participants received 6 mg of MK-0616 orally once daily (QD) for 8 weeks
- MK-0616 12 mg: Participants received 12 mg of MK-0616 orally QD for 8 weeks
- MK-0616 18 mg: Participants received 18 mg of MK-0616 orally QD for 8 weeks
- MK-0616 30 mg: Participants received 30 mg of MK-0616 orally QD for 8 weeks
- Placebo: Participants received MK-0616-matching placebo orally QD for 8 weeks
Period: Overall Study
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
Started | 77 | 76 | 76 | 76 | 76
Treated | 77 | 76 | 76 | 76 | 75
Completed | 75 | 76 | 74 | 74 | 74
Not Completed | 2 | 0 | 2 | 2 | 2
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0
Not completed — Not Recorded | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-0616 6 mg: Participants received 6 mg of MK-0616 orally QD for 8 weeks
- Total: Total of all reporting groups
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo | Total
Number analyzed (Participants) | 77 | 76 | 76 | 76 | 76 | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (10.3) | 62.0 (9.4) | 62.0 (9.2) | 60.9 (10.2) | 60.6 (9.3) | 61.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 39 | 38 | 38 | 188
  Male | 39 | 41 | 37 | 38 | 38 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 29 | 31 | 31 | 37 | 154
  Not Hispanic or Latino | 51 | 46 | 45 | 45 | 38 | 225
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 5 | 2 | 5 | 21
  Asian | 18 | 13 | 11 | 13 | 8 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 2 | 9 | 4 | 24
  White | 49 | 48 | 55 | 44 | 54 | 250
  More than one race | 2 | 5 | 3 | 8 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Randomization Strata: Background Statin Dose [Count of Participants; unit: Participants] — Participants were stratified by the following background statin dose: no statin therapy, low-intensity to moderate-intensity statin therapy, or high-intensity statin therapy.
  Participants
    No Statin Therapy | 30 | 29 | 31 | 30 | 30 | 150
    Low- to Moderate-intensity Statin Therapy | 27 | 27 | 26 | 26 | 26 | 132
    High-intensity Statin Therapy | 20 | 20 | 19 | 20 | 20 | 99
Randomization Strata: Renal Function [Count of Participants; unit: Participants] — Estimated glomerular filtration rate (eGFR) was calculated using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine. Participants were stratified by the following renal function at baseline: eGFR ≥60 vs <60 ml/min/1.73 m^2.
  Participants
    eGFR ≥60 ml/min/1.73 m^2 | 71 | 72 | 72 | 71 | 71 | 357
    eGFR <60 ml/min/1.73 m^2 | 6 | 4 | 4 | 5 | 5 | 24
Baseline Low-density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — Blood samples were taken at baseline to determine baseline LDL-C levels.
  mg/dL | 116.5 (37.0) | 117.3 (36.4) | 123.7 (35.1) | 119.4 (36.7) | 120.7 (28.3) | 119.5 (34.8)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 8
Description: Blood samples were collected at baseline and after 8 weeks of treatment to assess mean percent change in LDL-C. Based on a constrained longitudinal analysis (cLDA) model including terms for treatment, time, baseline statin intensity, baseline renal function, and the interaction of treatment by time. The percent change from baseline in LDL-C at week 8 was reported.
Time Frame: Baseline and up to Week 8
Population: All randomized participants who received at least one dose of study intervention, had at least one observation for the analysis endpoint, and had baseline data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
Number analyzed (Participants) | 75 | 75 | 74 | 73 | 72
Percentage Change | -40.0 [-45.2 to -34.8] | -54.5 [-59.8 to -49.2] | -57.9 [-63.2 to -52.6] | -59.7 [-65.0 to -54.5] | 1.2 [-4.1 to 6.5]
Statistical Analysis 1: Comparison: MK-0616 6 mg vs Placebo; Test type: Superiority — One-sided p-value and difference in least squares means based on a cLDA model including terms for treatment, time, baseline statin intensity, baseline renal function, and the interaction of treatment by time; p < 0.001, cLDA; Difference in Least Squares Means = -41.2, 95% CI 2-sided [-47.8 to -34.7] — MK-0616 6 mg minus Placebo
Statistical Analysis 2: Comparison: MK-0616 12 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -55.7, 95% CI 2-sided [-62.3 to -49.1] — MK-0616 12 mg minus Placebo
Statistical Analysis 3: Comparison: MK-0616 18 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -59.1, 95% CI 2-sided [-65.7 to -52.5] — MK-0616 18 mg minus Placebo
Statistical Analysis 4: Comparison: MK-0616 30 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -60.9, 95% CI 2-sided [-67.6 to -54.3] — MK-0616 30 mg minus Placebo

2. Primary Outcome: Percentage of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced at least one AE was reported.
Time Frame: Up to approximately 17 Weeks
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
Number analyzed (Participants) | 77 | 76 | 76 | 76 | 75
Percentage of Participants | 44.2 | 39.5 | 43.4 | 42.1 | 44.0
Statistical Analysis 1: Comparison: MK-0616 6 mg vs Placebo; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in Percentage = 0.2, 95% CI 2-sided [-15.5 to 15.8] — MK-0616 6 mg minus Placebo
Statistical Analysis 2: Comparison: MK-0616 12 mg vs Placebo; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in Percentage = -4.5, 95% CI 2-sided [-20.0 to 11.2] — MK-0616 12 mg vs Placebo
Statistical Analysis 3: Comparison: MK-0616 18 mg vs Placebo; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in Percentage = -0.6, 95% CI 2-sided [-16.3 to 15.1] — MK-0616 18 mg vs Placebo
Statistical Analysis 4: Comparison: MK-0616 30 mg vs Placebo; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in Percentage = -1.9, 95% CI 2-sided [-17.5 to 13.8] — MK-0616 30 mg minus Placebo

3. Primary Outcome: Percentage of Participants Who Discontinued Study Intervention Due to AEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinued study intervention due to AEs was reported.
Time Frame: Up to approximately 9 Weeks
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
Number analyzed (Participants) | 77 | 76 | 76 | 76 | 75
Percentage of Participants | 2.6 | 0.0 | 2.6 | 2.6 | 1.3

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Week 8
Description: Blood samples were collected at baseline and after 8 weeks of treatment to assess mean percent change in ApoB. The least square mean and 95% CI were obtained from fitting a cLDA model including terms for treatment, time, baseline statin intensity, baseline renal function, and the interaction of treatment by time. The percent change from baseline in ApoB at week 8 was reported.
Time Frame: Baseline and up to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
Number analyzed (Participants) | 76 | 75 | 74 | 74 | 72
Percentage Change | -32.8 [-37.6 to -27.9] | -45.8 [-50.7 to -40.9] | -48.7 [-53.6 to -43.8] | -51.8 [-56.7 to -47.0] | 0.0 [-4.9 to 4.9]
Statistical Analysis 1: Comparison: MK-0616 6 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -32.8, 95% CI 2-sided [-38.6 to -26.9] — MK-0616 6 mg minus Placebo
Statistical Analysis 2: Comparison: MK-0616 12 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -45.8, 95% CI 2-sided [-51.7 to -39.9] — MK-0616 12 mg minus Placebo
Statistical Analysis 3: Comparison: MK-0616 18 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -48.7, 95% CI 2-sided [-54.6 to -42.8] — MK-0616 18 mg minus Placebo
Statistical Analysis 4: Comparison: MK-0616 30 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Square Means = -51.8, 95% CI 2-sided [-57.7 to -45.9] — MK-0616 30 mg minus Placebo

5. Secondary Outcome: Percent Change From Baseline in Non-High-density Lipoprotein Cholesterol (Non-HDL-C) at Week 8
Description: Blood samples were collected at baseline and after 8 weeks of treatment to assess mean percent change in non-HDL-C. The least square mean and 95% CI were obtained from fitting a cLDA model including terms for treatment, time, baseline statin intensity, baseline renal function, and the interaction of treatment by time. The percent change from baseline in non-HDL-C at week 8 was reported.
Time Frame: Baseline and up to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
Number analyzed (Participants) | 74 | 76 | 74 | 73 | 72
Percentage Change | -34.4 [-39.6 to -29.2] | -49.0 [-54.3 to -43.7] | -51.8 [-57.1 to -46.4] | -54.3 [-59.6 to -49.1] | 1.5 [-3.9 to 6.8]
Statistical Analysis 1: Comparison: MK-0616 6 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -35.9, 95% CI 2-sided [-42.4 to -29.4] — MK-0616 6 mg minus Placebo
Statistical Analysis 2: Comparison: MK-0616 12 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -50.5, 95% CI 2-sided [-57.0 to -44.0] — MK-0616 12 mg minus Placebo
Statistical Analysis 3: Comparison: MK-0616 18 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -53.2, 95% CI 2-sided [-59.7 to -46.7] — MK-0616 18 mg minus Placebo
Statistical Analysis 4: Comparison: MK-0616 30 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, cLDA; Difference in Least Squares Means = -55.8, 95% CI 2-sided [-62.3 to -49.3] — MK-0616 30 mg minus Placebo

6. Secondary Outcome: Percentage of Participants With LDL-C Value at Goal at Week 8
Description: LDL-C goal was defined as: LDL-C <70 mg/dL (<1.81 mmol/L) in participants with clinical atherosclerotic cardiovascular disease (ASCVD), LDL-C <100 mg/dL (<2.59 mmol/L) in participants with an ASCVD risk-equivalent and/or a 10-year risk of having an ASCVD event that is ≥7.5%, OR LDL-C <130 mg/dL (<3.37mmol/L) in participants with a 10-year risk of having an ASCVD event that is ≥5.0% and <7.5%. The percentage of participants with LDL-C value at goal at week 8 were reported.
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study intervention and had at least one observation for the analysis endpoint were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
Number analyzed (Participants) | 77 | 76 | 76 | 76 | 75
Percentage of Participants | 80.5 | 85.5 | 90.8 | 90.8 | 9.3
Statistical Analysis 1: Comparison: MK-0616 6 mg vs Placebo; Test type: Superiority — One-sided p-value and difference in percentage based on Miettinen & Nurminen method, with sample size weighting, stratified by background statin intensity; p < 0.001, Miettinen & Nurminen; Difference in Percentage = 69.2, 95% CI 2-sided [56.2 to 79.0] — MK-0616 6 mg minus Placebo
Statistical Analysis 2: Comparison: MK-0616 12 mg vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Difference in Percentage = 75.2, 95% CI 2-sided [62.9 to 84.0] — MK-0616 12 mg minus Placebo
Statistical Analysis 3: Comparison: MK-0616 18 mg vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Difference in Percentage = 79.2, 95% CI 2-sided [67.1 to 87.1] — MK-0616 18 mg minus Placebo
Statistical Analysis 4: Comparison: MK-0616 30 mg vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Difference in Percentage = 79.5, 95% CI 2-sided [67.9 to 87.4] — MK-0616 30 mg minus Placebo

ADVERSE EVENTS:
Time Frame: Up to approximately 17 weeks
Description: The population analyzed for the All-Cause Mortality was all randomized participants. The population analyzed for AEs was all randomized participants who received at least one dose of study treatment, corresponding to the study treatment they actually received.
Arm/Group | MK-0616 6 mg | MK-0616 12 mg | MK-0616 18 mg | MK-0616 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/76 | 1/76 | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/77 | 3/76 | 2/76 | 2/76 | 0/75
Other Adverse Events (participants affected / at risk) | 11/77 | 13/76 | 15/76 | 8/76 | 15/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0616 6 mg (N=77) | MK-0616 12 mg (N=76) | MK-0616 18 mg (N=76) | MK-0616 30 mg (N=76) | Placebo (N=75)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0616 6 mg (N=77) | MK-0616 12 mg (N=76) | MK-0616 18 mg (N=76) | MK-0616 30 mg (N=76) | Placebo (N=75)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 5 (5)
COVID-19 (Infections and infestations) | 6 (6) | 1 (1) | 5 (5) | 4 (4) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT05261126/Prot_SAP_000.pdf